CLINICAL TRIAL: NCT05351879
Title: A Phase I/II Open Label Pilot Study to Evaluate the Safety and Feasibility of an Additional Intralymphatic Booster Administration of GAD-alum (Diamyd®) in Individuals With Type 1 Diabetes
Brief Title: Evaluation of a Booster Administration of GAD-alum (Diamyd®) in Individuals With Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Diamyd Medical AB (Industry)
Responsible Party: Principal Investigator, Johnny Ludvigsson, MD, PhD, Professor, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAGNODE-B
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diamyd; Diabetes; Diabetes Type 1; Type 1 Diabetes; Type 1 Diabetes Mellitus; GAD65; GAD-Alum; rhGAD65 (Recombinant Human GAD with molecular mass 65,000); Vitamin D; Diabetes mellitus Type 1; Glutamic acid decarboxylase
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GAD-Alum (DIamyd) 40 μg/mL and Vitamin D (Experimental): Patients with a Vitamin D level <100 nmol/L (40 ng/mL) at screening will receive oral Vitamin D supplementation (2000 IU daily) for 60 days, starting 30 days prior to the injection.
  On Visit 2 (Day 0), patients eligible for the study will receive one intralymphatic injection of 4µg Diamyd.
  Interventions: Biological: GAD-alum (Diamyd) 40 μg/mL

INTERVENTIONS:
Biological: GAD-alum (Diamyd) 40 μg/mL — Recombinant Human Glutamic Acid Decarboxylase (rhGAD65) adsorbed to Alhydrogel at a concentration of 40 μg/mL and is given as a sterile solution for intralymphatic injection

SUMMARY:
The objective of the study is to evaluate the feasibility and safety of administering a 4th or 5th intralymphatic booster dose of GAD-alum (Diamyd®) to T1D patients carrying HLA DR3-DQ2, who have earlier been treated with three or four intralymphatic doses of GAD-alum (Diamyd®) respectively.

DETAILED DESCRIPTION:
The study is a phase I/II, single arm, open label pilot clinical trial. Eligible patients will receive one booster injection of Diamyd® administered into an inguinal lymph node.

The patients will be assessed for eligibility at the screening visit (Visit 1). Patients with a Vitamin D level <100 nmol/L (40 ng/mL) at screening will receive oral Vitamin D supplementation (2000 IU daily) for 60 days, starting 30 days prior to the injection. On Visit 2 (Day 0), patients eligible for the study will receive one intralymphatic injection of 4µg Diamyd®

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent given by patients and/or patient's parent(s) or legal acceptable representative(s) (guardian(s)) according to national regulations
2. T1D according to the ADA classification
3. Carry HLA DR3-DQ2 haplotype
4. Prior participation in either the DIAGNODE-1 or the DIAGNODE-2, having received four or three intralymphatic injections of Diamyd, respectively.
5. Females must agree to avoid pregnancy and have a negative urine pregnancy test.

Patients of childbearing potential must agree to use adequate contraception, until 90 days after the administration of Diamyd. Adequate contraception is as follows:

For females of childbearing potential:

1. oral (except low-dose gestagen (lynestrenol and norestisteron)), injectable, or implanted hormonal contraceptives
2. combined (estrogen and progestogen containing)
3. oral, intravaginal or transdermal progesterone hormonal contraception associated with inhibition of ovulation
4. intrauterine device
5. intrauterine hormone-releasing system (for example, progestin-releasing coil)
6. bilateral tubal occlusion
7. vasectomized male (with appropriate post vasectomy documentation of the absence of sperm in the ejaculate)
8. male partner using condom
9. abstinence from heterosexual intercourse

For males of childbearing potential:

1. condom (male)
2. abstinence from heterosexual intercourse

Exclusion Criteria:

1. Previous or current treatment with immunosuppressant therapy (although topical or inhaled steroids are accepted)
2. Continuous treatment with anti-inflammatory drug (sporadic treatment e.g. because of headache or in connection with fever a few days will be accepted)
3. Treatment with any oral or injected anti-diabetic medications other than insulin
4. Treatment with Vitamin D, marketed or not, or unwilling to abstain from such medication during the supplementation period
5. A history of anemia or significantly abnormal hematology results at screening
6. A history of epilepsy, head trauma or cerebrovascular accident, or clinical features of continuous motor unit activity in proximal muscles
7. Clinically significant history of acute reaction to vaccines or other drugs in the past, including Diamyd
8. Treatment with any vaccine, including influenza or Covid19 vaccine, within 1 month prior to planned study drug dose administration or planned treatment with any vaccine up to 1 month after the injection with study drug
9. Participation in clinical trials (other than DIAGNODE-1 and DIAGNODE-2) with a new chemical entity within the previous 3 months
10. Inability or unwillingness to comply with the provisions of this protocol
11. A history of alcohol or drug abuse
12. A significant illness other than diabetes within 2 weeks prior to first dosing s
13. Ongoing diagnosed or suspected post-Covid19 syndrome
14. Known HIV or hepatitis
15. Females who are lactating or pregnant (the possibility of pregnancy must be excluded by urine βHCG on-site within 24 hours prior to the Diamyd treatment)
16. Presence of associated serious disease or condition, including active skin infections that preclude intralymphatic injection, which in the opinion of the investigator makes the patient non-eligible for the study
17. Deemed by the investigator not being able to follow instructions and/or follow the study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Number of Clinically Significant Abnormal Results from Physical examinations, including neurological and Vital Signs assessments | 12 months
Injection site reactions | 3 months
Occurrence of AEs and SAEs | 12 months
Number of Clinically Significant Abnormal Results From Laboratory measurements (hematology, clinical chemistry) and Urine analysis. | 12 months

SECONDARY OUTCOMES:
Change in Stimulated C-peptide During a MMTT | Baseline and 12 months
Change in HbA1c | Baseline and 12 months
Change in daily exogenous insulin consumption | Baseline and 12 months
Change in insulin-dose-adjusted HbA1c (IDAA1c) | Baseline and 12 months
Change in time in glycemic target range 3.9 to 10 mmol/L | Baseline and 12 months
Change in time in hyperglycemic range > 10 mmol/L | Baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Ludvigsson, Professor, Principal Investigator — Linkoeping University
Locations (1):
- Kliniska Forskningsenheten (Hudmottagningen), Universitetssjukhuset Linköping, Linköping, Sweden